CLINICAL TRIAL: NCT05046574
Title: Integrating Animal-assisted Therapy in Stroke Rehabilitation: a Randomized Controlled Trial Assessing the Impact on Psychological State and Functional Recovery of Patients, as Well as Wellbeing of Therapy Dogs
Brief Title: A Study to Evaluate Animal-assisted Therapy in Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Purina Petcare (Unknown)
Responsible Party: Principal Investigator, Arya B. Mohabbat, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-005175
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy dog during stroke rehabilitative therapy sessions (Experimental): Participants randomized to this arm will have a therapy dog present during their stroke rehabilitative therapy sessions.
  Interventions: Other: Stroke rehabilitative therapy sessions with therapy dog present
- No therapy dog during stroke rehabilitative therapy sessions (No Intervention): Participants randomized to this arm will have stroke rehabilitative therapy sessions per standard of care with no therapy dog present.

INTERVENTIONS:
Other: Stroke rehabilitative therapy sessions with therapy dog present — Therapy dog will be present during stroke rehabilitative therapy sessions. This is expected to be at least three times a week per 7-day period.
  Arms: Therapy dog during stroke rehabilitative therapy sessions

SUMMARY:
The investigators hypothesize that the presence of a Mayo Clinic certified therapy dog will provide additional benefits above typical treatment for patients currently enrolled in the Mayo Clinic Stroke Rehabilitation Unit.

DETAILED DESCRIPTION:
The objectives of this study are to measure the effects of a therapy dog embedded in stroke rehabilitation sessions on the patients' functional recovery, depression, anxiety, motivation, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older.
* Patient must be in the comprehensive in-patient stroke rehabilitation program.
* Patient must have a stroke from any cause.
* Patients must be able and willing to give informed consent.
* Patients must be able to speak English as the questionnaires being used are only available in English.

Exclusion Criteria:

* Patient who has a pacemaker.
* Patient who is pregnant.
* Patient who is deemed inappropriate to the study by the medical professional.
* Patient who is unable to give informed consent.
* Patient who is unable to speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety | Baseline through inpatient stay, an average of 2 weeks.
  Change in anxiety from admission to discharge of hospital stay through use of the General Anxiety Disorder scale (GAD-7). GAD-7 scores range from 0 to 21 with higher scores indicating greater severity of anxiety.
Change in Depression | Baseline through inpatient stay, an average of 2 weeks.
  Change in depression from admission to discharge of hospital stay through the use of the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 scores range from 0 to 27 with higher scores indicating greater severity of depression.
Change in Quality of Life Outcomes | Baseline through inpatient stay, an average of 2 weeks.
  Change in quality of life outcomes from admission to discharge of hospital stay through the use of the Stroke Specific Quality of Life Scale (SSQLS). The SSQL has 49 items that covers 12 domains. The SSQL scores range from 49 to 245 with higher scores indicating a better health related quality of life.
Change in motivation | Baseline through inpatient stay, an average of 2 weeks.
  Change in motivation from admission to discharge of hospital stay through the use of the Pittsburgh Rehabilitation Participation Scale (PRRS). The PRRS is a clinician-rated instrument used to evaluate patients' participation in therapy. This questionnaire contains one item, asking therapists to rate the patient's effort and motivation during the therapy session based on a 6-point scale.
Change in overall functional recovery | Baseline through inpatient stay, an average of 2 weeks.
  Change in overall functional recovery from admission to discharge of hospital stay through the use of the Self-Care and Mobility Quality Measures (SMQM). The SMQM is a clinician-rated instrument used to measure self-care and mobility measures. The clinician rates each item on a 6-point scale. A higher domain score indicates that the patient has a better independency in the functional performance of that domain.

CONTACTS AND LOCATIONS:
Overall Officials: Arya Mohabbat, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials